CLINICAL TRIAL: NCT00832013
Title: Safe Administration of Propofol for Sedation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Anesthesiologists' Society (Other)
Responsible Party: Dr. Mark Ansermino, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H07-02846
Record Dates: First submitted 2009-01-27; First posted 2009-01-29 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Sedation
Keywords: Propofol; sedation; pediatric; Induction of sedation
MeSH Terms: interventions — Propofol

ARMS (2):
- 1 (Active Comparator): Propofol 1 % at a dose of 4mg/kg will be administered intravenously via a standard Medex Protégé® 3010 (Medex-A Furon. Healthcare Company, Duluth, GA, USA) infusion pump at a constant rate determined by the randomization schedule. Fresh gas flow will be maintained at 6 l/min throughout the induction procedure with the FiO2 increased to 0.5. Full cardiovascular, respiratory and EEG monitoring will continue during induction of anesthesia.
  Once the loading dose of propofol has been delivered the propofol infusion will be maintained at a rate of 200mcg/kg/min or as determined by the attending anesthesiologist whilst the end-point respiratory responses are observed.
  Interventions: Drug: Propofol
- 2 (Active Comparator): Same procedure as above. These subjects will be stratified by age and randomized, using the Biased Coin Design (BCD) principle to determine the infusion rate of propofol for delivery of the induction dose.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — See detailed description
  Arms: 1
Drug: Propofol — See detailed description
  Arms: 2

SUMMARY:
Advances in health care require that more children are given sedation to allow doctors to perform investigations or minor procedures. Sedation drugs have traditionally been given orally (swallowed) by children. However, oral sedation drugs have unpredictable characteristics, such as duration of sedation, which may result in difficulties performing the planned procedure.

Anesthetic drugs are now invariably used for sedation in children. These are given through an IV (skinny plastic tube inserted in to a vein). Propofol (white liquid) is the anesthetic drug most commonly used for sedation at BC Children's Hospital for sedation. Propofol has several advantages, including an accurately controllable depth of sedation (how deeply asleep), minimal effect on the heart and circulation and control of reflexes (e,g coughing) during the procedure. Propofol also promotes rapid recovery with less sickness and an earlier return to normal functioning following the procedure.

While propofol has many advantages it can cause respiratory depression (reduced breathing rate). This reduction in breathing is more common if propofol is given quickly. When your child is given propofol for their proposed procedure this is performed by a pediatric anesthesiologist who is skilled in supporting breathing should this be required. If your child does not participate in this study they will still receive propofol administered by the anesthesiologist as this is our usual practice. It would be routine to administer the propofol rapidly and then support breathing for a few minutes. This is very safe in the hands of an expert anesthesiologist but can be sometimes more risky in other settings where extensive monitoring and anesthesiologists are not available. This is the setting that propofol is used in many institutions.

Our goal is to determine how quickly propofol can be given without reducing breathing to the point that help with breathing is required.

DETAILED DESCRIPTION:
Purpose Advances in minimally invasive radiological and surgical techniques demand that increasing numbers of children are given sedation or anesthesia to facilitate these procedures, frequently performed on an out-patient or day-care basis. Most are performed outside the operating room environment, with intensivists and emergency physicians administering over 55 % of sedation episodes, and only 19% being performed by anesthesiologists in North America. It is well documented that risks of complications during sedation exceed those experienced during the much more controlled environment of general anesthesia, with a twelve-fold increased risk of mortality when sedation is administered outside the operating room.

Sedative agents have traditionally been administered orally to children. However, characteristics of oral sedation drugs, such as unpredictable depth and duration of sedation resulting from variable drug absorption and prolonged duration of drug effect, have resulted in both high failure and complication rates. Recently, intravenous (IV) anesthetic drugs with more accurately titratable and predictable characteristics have gained popularity for a variety of sedation procedures. Propofol is the most commonly used intravenous agent for these procedures in North America.

Hypothesis The maximum safe infusion rate for an induction dose of propofol administered to children for sedation can be reliably predicted. Safety will be optimized by preventing apnoea whilst minimizing the time for induction of sedation and ensuring an adequate depth of sedation is achieved.

Justification Propofol is an intravenous (IV) anesthetic agent used for induction and maintenance of anesthesia in both adults and children. Propofol has several characteristics favouring its use, including an accurately titratable depth of anesthesia, cardiovascular stability, suppression of upper airway reflexes, rapid recovery with reduced post-operative nausea and vomiting and overall earlier return to pre-anesthetic functional state. At lower doses, propofol may also be used to maintain a level of sedation for radiological imaging or endoscopic investigations.

While propofol provides many advantages it does cause significant respiratory depression. Adverse respiratory events have been reported to be similar in both adults and children. Propofol induced respiratory depression may lead to hypoxemia requiring the provision of supplemental oxygen by mask and/or manual positive pressure ventilation.8 Artificial ventilation requires significant expertise and if poorly managed may result in gastric insufflation, pulmonary aspiration or hypoxia, all of which can lead to devastating complications such as permanent brain injury or death. The maximum dose or rate of administration of propofol that causes respiratory depression in children has yet to be accurately defined. Age specific effects have also not been reported.

Objectives

Primary aim:

•Develop a safe dosing schedule for propofol administration in children that will ensure spontaneous ventilation is maintained in at least 95% of subjects.

Secondary aim:

•Model the effects of propofol induction administered by intravenous infusion to facilitate the prediction of dosing schedules for different doses, different end-points in different clinical scenarios.

Research Method Prospective randomized study. Subjects will be randomly assigned to receive a predetermined infusion rate for propofol during induction of sedation.

Statistical Analysis A graphical representation of each data point with crossovers will be produced. Data will be analysed on a per protocol basis using the pooled-adjacent-violators algorithm to estimate the maximal infusion rate whilst preserving spontaneous ventilation. We will apply the boot-strap methods implemented by Pace to compute 95 % confidence limits. The effect of age, will be assessed by performing separate analyses in the age-strata.

To model the ventilatory effects of propofol, we will develop a mathematical model of human respiratory control. We will base this on the respiratory model proposed by Ursino (Ursino Model)19-21 which is a three compartment model comprising the lung, brain and tissues for gas exchange. We will enhance the model to include ventilatory regulation, along with pharmacokinetic and pharmacodynamic models of propofol including a respiratory effect site. The identification of suitable parameters for the model will include non-linear fitting of the clinical data (age, weight, BSA, ventilatory volumes, CO2 excretion, respiratory rate, and entropy).

ELIGIBILITY:
Inclusion Criteria:

All ASA category 1 and 2 children aged 6-15y for elective upper or lower gastrointestinal endoscopic investigations to be performed under sedation. Stratification by age (<9y, 9-12y, >12y) will be performed to ensure balanced allocation of age groups and allow for identification of age and weight specific effects.

Exclusion Criteria:

* Subjects with a history or signs of chronic lung disease;
* Active upper respiratory tract infection;
* Chronic opioid or other sedative drug therapy;
* Anticipated difficult airway, reflux, delayed gastric emptying;
* Other indications for endotracheal intubation;
* Subjects outwith the 5th or 95th centile of weight for age: translates to a minimum weight of 12kg at 3 years and maximum of 79kg at 15y.
* Contra-indications to propofol or lidocaine.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Positive result: Spontaneous ventilation continues following administration of the full loading dose of propofol by infusion. | Before and during surgery

SECONDARY OUTCOMES:
Negative result: Apnoea occurs (no breath for 20 seconds or oxygen saturation less than 90%) before the complete dose is administered or within 4 minutes of the end of the dose. | Before and during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ansermino, MD, Principal Investigator — University of British Columbia; Jon McCormack, Study Director — University of British Columbia; Eleanor Reimer, Study Director — University of British Columbia; Guy Dumont, Study Director — University of British Columbia; Prasad Shrawane, Study Director — University of British Columbia; Rollin Brant, Study Director — University of British Columbia
Locations (1):
- BC Children's Hospital, Department of Anesthesia, Vancouver, British Columbia, Canada